CLINICAL TRIAL: NCT02390674
Title: Evaluating the Effectiveness of Intravenous Ciclosporin on Reducing Reperfusion Injury in Patients Undergoing Primary Percutaneous Intervention: a Double-blind Randomised Controlled Trial
Brief Title: Ciclosporin to Reduce Reperfusion Injury in Primary PCI
Acronym: CAPRI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R&D 6327; 2014-002628-29 (EudraCT Number); BH120771 (Other Grant/Funding Number: NIHR BRC); 14/NE/1070 (Other: NRES Committee North East - Newcastle & North Tyneside 2)
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Myocardial Reperfusion Injury
MeSH Terms: conditions — Myocardial Reperfusion Injury | interventions — Cyclosporine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ciclosporin (Active Comparator): Single intravenous administration of ciclosporin (2.5mg per kilogram body weight) immediately prior to reperfusion during primary percutaneous coronary intervention. Ciclosporin is dissolved in saline (maximum concentration 2.5mg per millilitre)
  Interventions: Drug: Ciclosporin
- Saline (Placebo Comparator): Single intravenous administration of placebo (saline) immediately prior to reperfusion during primary percutaneous coronary intervention
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ciclosporin — Comparison between ciclosporin and placebo
  Other Names: Sandimmun
  Arms: Ciclosporin
Drug: Saline
  Arms: Saline

SUMMARY:
Routine primary percutaneous coronary intervention (PPCI) for a heart attack involves opening a blocked artery with a balloon then inserting a metal scaffold (stent) to hold the artery open. During this procedure inflammation can occur causing further damage to the heart. The objective of this trial is to determine whether administration of the drug ciclosporin prior to PPCI reduces the amount of damage to the heart relative to treatment with placebo. The damage to the heart is assessed after 12 weeks by an magnetic resonance imaging (MRI) scan. Patients are followed-up after 12 months participation in the study.

This is a single centre study looking to recruit 68 patients.

DETAILED DESCRIPTION:
Coronary heart disease is a condition in which the supply of blood and oxygen to the heart is reduced due to the narrowing of the arteries supplying the heart. A heart attack is caused when one of these arteries becomes blocked. Modern treatment for a heart attack is called primary percutaneous coronary intervention (PPCI). PPCI involves opening the blocked artery with a balloon and placing a stent (a small metal tube) in the artery to hold it open.

Research has shown that after opening the blocked artery, inflammation develops within the heart. This inflammation is generated by the immune system. Initial studies have suggested that certain immune system cells (T-cells) may be involved in causing much of the damage that occurs in the heart following a heart attack. The drug ciclosporin temporarily inhibits the immune system and it has been shown in a small number of patients that it reduces the size of the heart attack. The aim of this clinical trial is to investigate in a larger number of patients whether the size of the heart attack is reduced in patients treated with the drug ciclosporin prior to PPCI relative to patients treated with a placebo (saline).

To participate in the trial you must be having a large heart attack (STEMI - ST segment elevation myocardial infarction) and be undergoing a PPCI to unblock your artery. You must also be aged over 18 years. You will be randomised to receive either a single dose of the drug ciclosporin or placebo before your blocked artery is opened. Half the people will get the drug ciclosporin. This randomisation will enable us to compare the results to see whether treatment with ciclosporin reduces the size of the heart attack compared with placebo.

There may be no immediate benefit from taking part in the trial but the information we get from this trial will help improve the treatment of people having a heart attack in the future. As far as we know there are no disadvantages of taking part in the trial. If you are randomised to the 'drug' group, there is a very small risk of side effects from ciclosporin, such as high blood pressure and slight worsening of kidney function. We do not expect any side effects as the ciclosporin is only given once in the trial. On rare occasions allergic reactions have been observed. If any ciclosporin-related side effects were to occur, they would be expected soon after the drug was administered.

This is a single centre, randomised, double-blind, parallel group, placebo-controlled phase II/III trial comparing the efficacy of ciclosporin versus placebo in 68 patients with acute myocardial infarction undergoing PPCI. The trial is set in a tertiary care centre (Freeman Hospital, Newcastle upon Tyne, UK) and patients will be recruited over a period of 18 months. The trial is designed to show superiority regarding its primary endpoint. During initial hospitalisation following myocardial infarction, treatment is given once prior to performing the PPCI in the catheter laboratory. The duration of study for each patient is 12 months until final follow-up (12 weeks randomised controlled trial (RCT) followed by 9 months study follow-up). Should treatment with ciclosporin look promising, a larger trial will be designed to evaluate ciclosporin treatment fully. In contrast to the previous study, this trial is not restricted to anterior STEMI patients. It will also analyse changes in inflammatory response following reperfusion and will use MRI (current gold standard) in every patient to quantify infarct size, ejection fraction and microvascular obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with acute myocardial infarction (STEMI) and undergoing primary percutaneous coronary intervention (PPCI)
* Age above 18 years
* Presenting within 6 hours of the onset chest pain and ST segment elevation. The culprit coronary artery has to be a major coronary artery with a diameter of at least 3mm and has to be proximally occluded (TIMI flow grade 0-1) at the time of admission coronary angiography

Exclusion Criteria:

* Patients with any disorder associated with immunological dysfunction (acute or chronic inflammatory or neoplastic co-existing disease, known positive serology for HIV, or hepatitis)
* Clinically unstable patients (haemodynamically unstable, cardiogenic shock, unconscious patients)
* Patients with evidence of coronary collaterals to the infarct area
* Patients with an open (TIMI > 1) culprit coronary artery at the time of angiography.
* Previous myocardial infarction
* Previous thrombolytic therapy
* Patients with known hypersensitivity to ciclosporin or to egg, peanut or soya-bean proteins.
* Patients with known renal insufficiency (either known glomerular filtration rate (GFR) <30 ml/min/1.73m2) or current medical care for severe renal insufficiency.
* Known liver insufficiency
* Uncontrolled hypertension (>180/110 mmHg)
* Patients treated with any compound containing hypericum perforatum, stiripentol, Aliskiren, Bosentan or Rosuvastatin or with an active treatment that might modify blood concentration of ciclosporin.
* Female patients currently pregnant or women of childbearing age who are not using contraception (verbal diagnosis). Female patients of childbearing potential who are using contraception but are subsequently found to have a positive urine pregnancy test (pregnancy test performed as soon as reasonably practicable after investigational medicinal product (IMP) administration).
* Contraindication to cardiac MRI:

  * Pacemaker
  * Implantable defibrillator
* Patients unable to undergo cardiac MRI for any of the following reasons:

  * Frailty - as judged by the clinician. Frailty is defined as meeting three out of the five following criteria: low grip strength, low energy, slowed walking speed, low physical activity and/or unintentional weight loss. Due to the tight time constraints and emergency setting of this trial the clinician cannot test all these parameters and will need to exercise their judgment.
  * Claustrophobic - patients who cannot take elevators or who are afraid of narrow or enclosed spaces.
  * Breathlessness - patients who suffer from breathlessness at rest or low exercise level (e.g. while walking on the level).
* Use of other investigational study drugs within 30 days prior to trial entry (defined as date of randomisation into trial). Co-enrolment with other studies is not allowed.
* Lack of capacity to give initial verbal consent
* Life expectancy <1year due to non-cardiac illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-03; Primary Completion 2017-04 (Actual); Study Completion 2017-11-11 (Actual)

PRIMARY OUTCOMES:
Change in infarct size | 12 weeks after primary percutaneous coronary intervention (PPCI)
  Change in infarct size 12 weeks post-PPCI as measured by cardiac MRI

SECONDARY OUTCOMES:
Change in microvascular obstruction | Measured once between day 2 and day 7 after PPCI
  Microvascular obstruction after 2-7 days as measured by a single cardiac MRI scan
Change in salvage index | Measured once between day 2 and day 7 after PPCI
  Salvage index after 2-7 days as measured by a single cardiac MRI scan
Change in T lymphocyte count | 5, 15, 30, 60 and 90 minutes
  Change in T lymphocyte counts relative to baseline at 5, 15, 30, 60 and 90 minutes post-reperfusion

CONTACTS AND LOCATIONS:
Overall Officials: Ioakim Spyridopoulos, PhD, MD, Principal Investigator — Newcastle University
Locations (1):
- Newcastle Clinical Trials Unit, Newcastle upon Tyne, Tyne and Wear, United Kingdom

REFERENCES:
- [Derived] Gatsiou A, Tual-Chalot S, Napoli M, Ortega-Gomez A, Regen T, Badolia R, Cesarini V, Garcia-Gonzalez C, Chevre R, Ciliberti G, Silvestre-Roig C, Martini M, Hoffmann J, Hamouche R, Visker JR, Diakos N, Wietelmann A, Silvestris DA, Georgiopoulos G, Moshfegh A, Schneider A, Chen W, Guenther S, Backs J, Kwak S, Selzman CH, Stamatelopoulos K, Rose-John S, Trautwein C, Spyridopoulos I, Braun T, Waisman A, Gallo A, Drakos SG, Dimmeler S, Sperandio M, Soehnlein O, Stellos K. The RNA editor ADAR2 promotes immune cell trafficking by enhancing endothelial responses to interleukin-6 during sterile inflammation. Immunity. 2023 May 9;56(5):979-997.e11. doi: 10.1016/j.immuni.2023.03.021. Epub 2023 Apr 25. PMID 37100060
- [Derived] Cormack S, Mohammed A, Panahi P, Das R, Steel AJ, Chadwick T, Bryant A, Egred M, Stellos K, Spyridopoulos I; CAPRI investigators. Effect of ciclosporin on safety, lymphocyte kinetics and left ventricular remodelling in acute myocardial infarction. Br J Clin Pharmacol. 2020 Jul;86(7):1387-1397. doi: 10.1111/bcp.14252. Epub 2020 Mar 11. PMID 32067256